CLINICAL TRIAL: NCT07011004
Title: Phase I Study of Cytokine Induced Memory-Like Natural Killer Cells Combined With Atezolizumb in Subjects With Relapsed or Refractory Acute Myelogenous Leukemia
Brief Title: A Study of Natural Killer Cells in Combination With Atezolizumab in People With Acute Myelogenous Leukemia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-356
Record Dates: First submitted 2025-05-30; First posted 2025-06-08 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Acute Myeloid Leukemia Refractory; Acute Myeloid Leukemia, in Relapse
Keywords: Atezolizumab; CIML-NK (Cytokine Induced Memory-Like Natural Killer Cells); 24-356
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Intervention Model Description: This is a phase I dose escalation and expansion study designed to evaluate the safety of cytokine induced, memory-like NK cells (CIML-NK) when combined with atezolizumab in patients with relapsed or refractory acute myelogenous leukemia (AML).
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cytokine Induced Memory-Like Natural Killer Cells Combined with Atezolizumb (Experimental): Pre-conditioning chemotherapy will consist of a standard lymphodepleting regimen including fludarabine 25 mg/m2 IV daily x 5 on days -6 to - 2 and cyclophosphamide 50 mg/kg IV x 2 on days -5 and -4 prior to the infusion of the CIML-NK cells. Standard MSKCC supportive care guidelines for infusion of chemotherapy including cyclophosphamide will be employed. On the day of infusion subjects will receive a single dose of atezolizumab IV over 60 minutes IV. Subjects will receive subcutaneous recombinant human IL-2 (rh-IL2) every other day x 6 doses beginning on day 0 via subcutaneous injection.
  Interventions: Biological: Cytokine Induced Memory-Like Natural Killer Cells; Biological: Atezolizumb; Biological: CIML-NK cell therapy

INTERVENTIONS:
Biological: Cytokine Induced Memory-Like Natural Killer Cells — Subjects will receive subcutaneous recombinant human IL-2 (rh-IL2) every other day x 6 doses beginning on day 0 via subcutaneous injection.
Biological: Atezolizumb — Single dose of Atezolizumab IV over 60 minutes IV.
Biological: CIML-NK cell therapy — CIML-NK cell therapy as an intravenous (IV) infusion

SUMMARY:
The researchers are doing this study is to find the highest dose of cytokine-induced memory-like (CIML) natural killer (NK) cells in combination with the drug atezolizumab that causes few or mild side effects in people with relapsed/refractory acute myelogenous leukemia (AML). The researchers will also look at whether the treatment combination works against participants' cancer.

ELIGIBILITY:
Inclusion Criteria:

Disease specific inclusion criteria:

* Subjects must have histologically confirmed acute myeloid leukemia that meets any of the following criteria:

  * Refractory to at least two attempts at prior induction therapy. An attempt is defined as either a single cycle of combination chemotherapy such as daunorubicin/anthracycline OR a single monthly cycle of a hypomethylating agent with venetoclax.
  * Patients with FLT3-ITD or -TKD mutations must have received at least one commercially available inhibitor of FLT3.
  * Patients with NPM1 mutation or rearrangements of MLL must be refractory to revumenib.
  * Patients with mutations in IDH1 or IDH2 must be refractory to at least one commercially available inhibitor of IDH1 or IDH2, respectively.
  * Relapsed AML when relapse occurred within 6 months of achieving an initial complete remission.
  * Patients must have either failed prior FDA approved agents or, in the opinion of the treating physician, have a sufficiently low probability of response to existing FDA approved agents to warrant treatment on an investigational protocol.

Other inclusion criteria:

* Patients aged 18 through 70 years old are eligible.
* Must have an available, haplotype mismatched related individual that meets criteria for cell donation according to the FACT guidelines.
* Patients must have Karnofsky performance status ≥70%.
* Adequate cardiac function as defined as a systolic LV ejection fraction ≥50% at rest and absence of New York Heart Association stage III or IV congestive heart failure.
* Adequate pulmonary function as defined as a resting SpO2 ≥ 92% on room air at rest.
* Serum bilirubin ≤ 5 mg/dL.
* AST and ALT ≤ 2.5x ULN unless thought to be disease related.
* Estimated or measured creatinine clearance > 50 mL/min.
* Subjects must be free from all systemic immune suppression for at least 4 weeks prior to the start of intended therapy.
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraception and agreement to refrain from donating eggs, as defined below: Women must remain abstinent or use contraceptive methods with a failure rate of <1% per year during the treatment period and for 5 months after the final dose of atezolizumab. Women must refrain from donating eggs during this same period.
* Negative HIV test at screening.
* Negative hepatitis B surface antigen (HBsAg) test at screening OR positive HBsAg is allowed if a negative HBcAb or a negative quantitative hepatitis B virus (HBV) (DNA < 500 IU/mL) assay are documented.
* Negative hepatitis C virus (HCV) antibody test at screening, or positive HCV antibody test followed by a negative HCV RNA test at screening The HCV RNA test must be performed for patients who have a positive HCV antibody test.
* For patients receiving therapeutic anticoagulation: Stable anticoagulant regimen for 2 weeks prior to enrollment.
* Timing of treatment relative to prior therapies:

  * Bridging therapy with hydrea is allowed but is required to be tapered off prior to NK infusion.
  * Any experimental biological treatments must be discontinued for at least 5 half-lives prior to initiation of study therapy.
  * Patients must be >5 half-lives from receipt of other cytotoxic or targeted therapy.

Exclusion Criteria:

* Prior allogeneic hematopoietic cell transplantation.
* Subjects with active/uncontrolled CNS leukemia. Subjects with prior CNS disease must have no detectable evidence of CSF disease for at least 4 weeks prior to enrollment.
* Subjects requiring systemic immunosuppression for any indication are excluded.
* Significant cardiovascular disease, as defined by:

  * New York Heart Association Class II or greater congestive heart failure.
  * Myocardial infarction, cerebrovascular accident, or other arterial vascular disease within 6 months prior to initiation of study treatment
  * Unstable arrhythmia
  * Unstable angina
* Subjects with isolated extramedullary disease without evidence of bone marrow involvement by immunohistochemistry.
* Female patients who are pregnant or breast-feeding or intend to become pregnant during study treatment or within 5 months after the final dose of atezolizumab. Women of childbearing potential must have a negative serum pregnancy test result within 14 days prior to initiation of study treatment with atezolizumab.
* Severe or uncontrolled infection prior to initiation of study treatment.
* Treatment with therapeutic oral or IV antibiotics within 2 weeks prior to initiation of study treatment, excluding prophylactic antimicrobial agents.
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan.
* Uncontrolled or symptomatic hypercalcemia (ionized calcium > 1.5 mmol/L, calcium >12 mg/dL, or corrected calcium greater than ULN)
* Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, anti-phospholipid antibody syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, or multiple sclerosis, with the following exceptions:

  * Patients with a history of autoimmune-related hypothyroidism who are on thyroid-replacement hormone are eligible for the study.
  * Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study.
  * Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all following conditions are met:

    * Rash must cover < 10% of body surface area.
    * Disease is well controlled at baseline and requires only low-potency topical corticosteroids.
    * There has been no occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high-potency or oral corticosteroids within the previous 12 months.
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently)
* Persons who do not meet the age and organ function criteria specified above.
* History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins
* Known hypersensitivity to Chinese hamster ovary cell products or to any component of the atezolizumab formulation.

Donor Inclusion Criteria:

* Donors must be eligible for apheresis according to standard FACT guidelines.
* Donors must not have an HLA genotype reactive against anti-HLA antibodies in the recipient.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-05-30 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
The maximum tolerated dose (MTD) | 2 years
  of the combination of CIML-NK cells with atezolizumab in subjects with r/r-AML. The MTD is defined as the highest dose with an observed incidence of DLT in no more than one out of six patients treated at a particular dose level.

SECONDARY OUTCOMES:
The response rate (CR/CRi) | 2 years
  Disease response assessments will be according to the ELN2022 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Shaffer, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering at Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited protocol activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk - Commack (Limited protocol activities), Commack, New York
  - Memorial Sloan Kettering West Harrison (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activites), Rockville Centre, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org